CLINICAL TRIAL: NCT01113008
Title: Remote Ischemic Postconditioning. Can it Prevent Myocardial Injury During Percutaneous Coronary Intervention?
Brief Title: Remote Ischemic Postconditioning in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Victoria (Other)
Collaborators: FUNDACIÓN IMABIS (Unknown); Red Temática de Investigación Cooperativa en Enfermedades Cardiovasculares (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PI-0327/2008
Record Dates: First submitted 2010-04-26; First posted 2010-04-29 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Myocardial Reperfusion Injury
Keywords: Myocardial Reperfusion Injury/mortality; Coronary angioplasty; Reperfusion; Myocardial Reperfusion Injury/prevention & control
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote postcondtioning (Experimental): Patients assigned to remote ischemic postconditioning (randomized controlled trial)
  Interventions: Procedure: Remote ischemic postconditioning
- Control group (Placebo Comparator)
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Remote ischemic postconditioning — Patients assigned to remote ischemic postconditioning will undergo three 5-minute cycles of ischemia using a blood-pressure cuff at 200 mmHg, placed on the non-dominant arm, interrupted twice for 5 minutes with the cuff deflated
  Arms: Remote postcondtioning
Procedure: Control group — In the control group the procedure will be limited to placing a deflated blood-pressure cuff (pressure: 0 mmHg) for 25 minutes.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the phenomenon of remote ischemic post-conditioning in humans. The minor myocardial damage associated with percutaneous revascularization procedures may be attenuated by producing controlled ischemia in the arms immediately after carrying out these procedures (remote ischemic post-conditioning). The justification and design of this clinical trial has been reported: Cardiology. 2011;119(3):164-9.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) has taken on an important role in the treatment of ischemic heart disease in recent years. However, the beneficial effects of revascularization are partly shadowed by post-reperfusion injury, which accounts for up to half the size of the reperfused myocardial infarct. Several drugs and procedures exist that might protect against this phenomenon. One of the most controversial of these strategies, which has shown promising results in experimental animal models, is remote ischemic post-conditioning. This involves inducing ischemia at a site remote from the heart after an ischemic coronary lesion to reduce the resulting myocardial infarct size.

The myocardial damage produced by ischemia-reperfusion associated with PCI is a known short- and long-term prognostic factor, and is associated with a greater risk of death, myocardial infarction and revascularization during the follow-up.

Our aim is to assess the phenomenon of remote ischemic post-conditioning in patients undergoing PCI, in whom the acute insult on the myocardium is determined by the angioplasty itself. Additionally, we aim to evaluate this phenomenon in a subgroup of diabetic patients, among whom the effectiveness of protective measures against post-reperfusion damage is more questioned.

We have designed a randomized, single-blinded interventional study involving 320 patients (40% diabetics) who are to undergo elective PCI. At the end of the angioplasty procedure, the patients assigned to remote ischemic post-conditioning will undergo three 5-minute cycles of ischemia using a blood-pressure cuff at 200 mmHg, placed on the non-dominant arm, interrupted twice for 5 minutes with the cuff deflated. In the control group the procedure will be limited to placing a deflated blood-pressure cuff (pressure: 0 mmHg) for 25 minutes.

The infarct size will be analyzed from an enzyme curve of troponin I and CK-MB values 0, 8, 16 and 24 hours after the procedure (primary endpoint). Measurements will also be taken of pH and lactate in the baseline sample (0 hours) and at 8 hours, and ultrasensitive C-reactive protein at 0 and 24 hours as a contrasted marker of inflammation in ischemic heart disease.

The follow-up, planned for one year, will seek to determine clinically interesting variables (secondary endpoint), such as readmission due to acute coronary syndrome, heart failure or major arrhythmic events and overall and cardiovascular mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing PCI due to stable angina
2. Patients undergoing PCI due to unstable angina
3. Patients undergoing PCI due NON Q acute myocardial infarction with normal troponin at inclusion moment (less than 1 ng/ml)

Exclusion Criteria:

1. Acute myocardial infarction during the previous two weeks
2. Chronic renal failure with baseline creatinine above 3 mg/dL

4. Collateral circulation of the revascularized artery (Rantrop >0) 5. Prior treatment with glibenclamide. 6. Inability to receive follow-up, blood test or lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel F Jiménez-Navarro, Doctor, Principal Investigator — Servicio Cardiología, Hospital Universitario Virgen de la Victoria
Locations (1):
- Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga, Spain

REFERENCES:
- [Background] JENNINGS RB, SOMMERS HM, SMYTH GA, FLACK HA, LINN H. Myocardial necrosis induced by temporary occlusion of a coronary artery in the dog. Arch Pathol. 1960 Jul;70:68-78. No abstract available. PMID 14407094
- [Background] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Jimenez-Navarro M, Gomez-Doblas JJ, Hernandez Garcia JM, Alonso-Briales J, Garcia Alcantara A, Gomez G, Rodriguez-Bailon I, de Teresa E. Does angina pectoris the week before protect against first acute myocardial infarction in patients with diabetes mellitus? Am J Cardiol. 2002 Jul 15;90(2):160-2. doi: 10.1016/s0002-9149(02)02442-6. No abstract available. PMID 12106849
- [Background] Iliodromitis EK, Kyrzopoulos S, Paraskevaidis IA, Kolocassides KG, Adamopoulos S, Karavolias G, Kremastinos DT. Increased C reactive protein and cardiac enzyme levels after coronary stent implantation. Is there protection by remote ischaemic preconditioning? Heart. 2006 Dec;92(12):1821-6. doi: 10.1136/hrt.2006.089060. Epub 2006 Jul 19. PMID 16855045
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Hoole SP, Heck PM, Sharples L, Khan SN, Duehmke R, Densem CG, Clarke SC, Shapiro LM, Schofield PM, O'Sullivan M, Dutka DP. Cardiac Remote Ischemic Preconditioning in Coronary Stenting (CRISP Stent) Study: a prospective, randomized control trial. Circulation. 2009 Feb 17;119(6):820-7. doi: 10.1161/CIRCULATIONAHA.108.809723. Epub 2009 Feb 2. PMID 19188504
- [Background] Staat P, Rioufol G, Piot C, Cottin Y, Cung TT, L'Huillier I, Aupetit JF, Bonnefoy E, Finet G, Andre-Fouet X, Ovize M. Postconditioning the human heart. Circulation. 2005 Oct 4;112(14):2143-8. doi: 10.1161/CIRCULATIONAHA.105.558122. Epub 2005 Sep 26. PMID 16186417
- [Background] Andreka G, Vertesaljai M, Szantho G, Font G, Piroth Z, Fontos G, Juhasz ED, Szekely L, Szelid Z, Turner MS, Ashrafian H, Frenneaux MP, Andreka P. Remote ischaemic postconditioning protects the heart during acute myocardial infarction in pigs. Heart. 2007 Jun;93(6):749-52. doi: 10.1136/hrt.2006.114504. Epub 2007 Apr 20. PMID 17449499
- [Background] Gritsopoulos G, Iliodromitis EK, Zoga A, Farmakis D, Demerouti E, Papalois A, Paraskevaidis IA, Kremastinos DT. Remote postconditioning is more potent than classic postconditioning in reducing the infarct size in anesthetized rabbits. Cardiovasc Drugs Ther. 2009 Jun;23(3):193-8. doi: 10.1007/s10557-009-6168-5. PMID 19255833
- [Derived] Carrasco-Chinchilla F, Munoz-Garcia AJ, Dominguez-Franco A, Millan-Vazquez G, Guerrero-Molina A, Ortiz-Garcia C, Enguix-Armada A, Alonso-Briales JH, Hernandez-Garcia JM, de Teresa-Galvan E, Jimenez-Navarro MF. Remote ischaemic postconditioning: does it protect against ischaemic damage in percutaneous coronary revascularisation? Randomised placebo-controlled clinical trial. Heart. 2013 Oct;99(19):1431-7. doi: 10.1136/heartjnl-2013-304172. Epub 2013 Jul 12. PMID 23850844

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Control group : In the control group the procedure will be limited to placing a deflated blood-pressure cuff (pressure: 0 mmHg) for 25 minutes.
- Remote Postcondtioning: Patients assigned to remote ischemic postconditioning (randomized controlled trial)
  Remote ischemic postconditioning : Patients assigned to remote ischemic postconditioning will undergo three 5-minute cycles of ischemia using a blood-pressure cuff at 200 mmHg, placed on the non-dominant arm, interrupted twice for 5 minutes with the cuff deflated
Period: Overall Study
Arm/Group | Control Group | Remote Postcondtioning
Started | 133 | 133
Completed | 133 | 133
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Postcondtioning | Control Group | Total
Number analyzed (Participants) | 118 | 114 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.1) | 64.4 (9.3) | 64.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 39 | 74
  Male | 83 | 75 | 158

OUTCOME MEASURES:

1. Primary Outcome: Maximum Increase of Troponin at 24 Hours
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Control Group | Remote Postcondtioning
Number analyzed (Participants) | 114 | 118
ng/ml | 0.478 [0.2839 to 0.6726] | 0.476 [0.2842 to 0.6686]

2. Secondary Outcome: Readmission Due to Acute Coronary Syndrome
Time Frame: 12 month
Measure: Number; unit: participants
Arm/Group | Control Group | Remote Postcondtioning
Number analyzed (Participants) | 133 | 133
participants | 1 | 4

3. Secondary Outcome: Cardiovascular Mortality
Time Frame: 12 month
Measure: Number; unit: participants
Arm/Group | Control Group | Remote Postcondtioning
Number analyzed (Participants) | 133 | 133
participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | Control Group | Remote Postcondtioning
Serious Adverse Events (participants affected / at risk) | 0/133 | 2/133
Other Adverse Events (participants affected / at risk) | 0/133 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=133) | Remote Postcondtioning (N=133)
Mortality (Cardiac disorders) | 0 (0) | 2 (2) — Mortality due to cardiovascular event in study follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No